CLINICAL TRIAL: NCT02854696
Title: Health Economic Analysis of Islet Cell Transplantation for Patients With Severe Forms of Brittle Type 1 Diabetes
Brief Title: Health Economic Analysis of Islet Cell Transplantation for the Stabilization of the Severe Forms of Type 1 Diabetes
Acronym: STABILOT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC14.453
Record Dates: First submitted 2016-03-04; First posted 2016-08-03 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Type 1 Diabetes
Keywords: Islet cell Transplantation; cost-effectiveness analysis; Cost-utility analysis; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Islet graft (Experimental): Patients who receive islet graft Intervention : Procedure/Surgery
  Interventions: Procedure: Islet graft
- Best medical care (Active Comparator): Patients who continue their optimal medical treatment (insulin pump therapy coupled with real time continuous glucose monitoring) Intervention : insulin treatment
  Interventions: Drug: best medical care

INTERVENTIONS:
Procedure: Islet graft — Patients will be transplanted with pancreatic islet cells
  Other Names: islet cell transplantation
  Arms: Islet graft
Drug: best medical care — Patients will continue their insulin treatment
  Other Names: insulin treatment
  Arms: Best medical care

SUMMARY:
The main goal is to perform a cost-utility analysis to compare islet cell transplantation versus best medical treatment (defined as Sensor augmented pump therapy) for patients with brittle type1 diabetes.

DETAILED DESCRIPTION:
The main goal is to perform a cost-utility analysis to compare islet cell transplantation versus best medical treatment (defined as Sensor augmented insulin pump therapy) for patients with brittle type1 diabetes.

ELIGIBILITY:
Inclusion Criteria :

* Suffering from diabetes since more than 5 years
* Patient with brittle type 1 diabetes despite an optimized insulin treatment and educational training will be included. A patient will be considered as experiencing a brittle type 1 diabetes if at least two criteria are present among: persistence of severe hypoglycemia, occurrence of ketoacidosis events without obvious etiology, diagnosis of unaware hypoglycemic episodes < 3 mmol/l based on CGM or self-monitoring blood glucose data, a mean blood glucose standard deviation>50%, MAGE index (Mean amplitude of glucose excursions)>60 mg/dl, LBGI index (low blood glucose index)>5, Clarke score≥4 or HYPOSCORE>800.
* Insulin needs < 0,85 U/kg/day
* HbA1c < 12% ;
* No residual insulin secretion (plasmatic basal and stimulated C-peptide < 0.3 ng/ml)
* Social Security membership or benefit from Social Security
* Patients who signed the consent form

Exclusion Criteria :

Exclusion criteria related to islet infusion:

* Hemostatic disorders, pre-existing liver disease (PAL, Gamma-GT, ASAT-ALAT >2N) or vesicular lithiasis.

Exclusion criteria related to diabetic complications:

* Evolutive proliferative retinopathy, evolutive nephropathy (Glomerular filtration rate <30 ml/min/1.73m2 and/or proteinuria >0.5g/day), evolutive cardiopathy or obliterative arteriopathy with trophic cutaneous lesions.

Exclusion criteria related to immunosuppressant use:

* Hemoglobin < 110mg/dL in women and < 120 mg/dL in men, leuconeutropenia, thrombopenia, systemic infection including chronic hepatitis B, C and VIH, neoplasia disease and hypertension>160/100 mmHg.
* Corticoid treatment (except for patient that benefited from a kidney graft with maintenance steroid therapy)
* Presence of anti-HLA antibody directed against the donor
* Positive B or T cells crossmatch

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incremental cost- utility ratio at 1 year | 1 year
  The primary endpoint will be the incremental cost-effectiveness ratio at one year for islet transplantation versus Best Medical Treatment of brittle type 1 diabetes.The effectiveness will be expressed as quality adjusted life years (QALYs) in a cost-utility analysis. QALYs are a composite measure of outcomes where utilities for health states (on 0-1 scale, where 0 corresponds to death and 1 to full health) act as qualitative weights to combine quantity and quality of life. The number of QALYs in each group will be assessed with the EuroQol 5 Dimensions questionnaire (EQ5D). The EQ-5D measures health status in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

SECONDARY OUTCOMES:
Cost-effectiveness ratio at 1 year | 1 year
  Assessment of the cost-effectiveness ratio at 1 year between islet cell transplantation versus best medical treatment (SAP therapy) for patients with brittle type 1 diabetes without impairment of vital prognosis. Two criteria of effectiveness will be used : the life years gained and the number of hypoglycemia
Assessment of individual medical benefit of quality of life | 6 months and 1year
  Evaluate with DQOL questionnaire
Assessment of individual medical benefit in terms of metabolic efficacy | 6 months and 1 year
  measured from the following criteria: severe hypoglycemia, HbA1c, stimulated C-peptide, fasting glucose, insulin dose or oral diabetes, glycemic variability
Assessment and comparison of individual medical benefit in terms of complications of islet cell transplantation between the two groups | 6 months and 1 year
  measured from in insulin independence, hospitalizations
Assessment and comparison of clinical benefit for patients with brittle type 1 diabetes with impairment of vital prognosis before and after islet cell transplantation | 1 year
  measured from DQOL, insulin independence, complications of islet cell transplantation
Assessment and comparison of costs for patients with brittle type 1 diabetes with impairment of vital prognosis before and after islet cell transplantation | 1 year
  measured from hospitalizations
Assessment of total cost of islet cell transplantation | 1 year
  Assessment of total cost of islet cell transplantation for patients with type 1 diabetes without impairment of vital prognosis, from pre-transplant period until 1 year after the last injection. Two perspectives will be used: French health care system and hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves BENHAMOU, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (11):
- France (10):
  - University Hospital of Besançon, Besançon
  - university hospital of Clermont Ferrand, Clermont-Ferrand
  - Grenoble University Hospital, Grenoble
  - University hospital of Lille, Lille
  - University Hospital of Lyon, Lyon
  - University Hospital of Montpellier, Montpellier
  - University hospital of Nancy, Nancy
  - university hospital of Nantes, Nantes
  - APHP, Paris
  - University hospital of Strasbourg, Strasbourg
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barton FB, Rickels MR, Alejandro R, Hering BJ, Wease S, Naziruddin B, Oberholzer J, Odorico JS, Garfinkel MR, Levy M, Pattou F, Berney T, Secchi A, Messinger S, Senior PA, Maffi P, Posselt A, Stock PG, Kaufman DB, Luo X, Kandeel F, Cagliero E, Turgeon NA, Witkowski P, Naji A, O'Connell PJ, Greenbaum C, Kudva YC, Brayman KL, Aull MJ, Larsen C, Kay TW, Fernandez LA, Vantyghem MC, Bellin M, Shapiro AM. Improvement in outcomes of clinical islet transplantation: 1999-2010. Diabetes Care. 2012 Jul;35(7):1436-45. doi: 10.2337/dc12-0063. PMID 22723582
- [Background] Beckwith J, Nyman JA, Flanagan B, Schrover R, Schuurman HJ. A health economic analysis of clinical islet transplantation. Clin Transplant. 2012 Jan-Feb;26(1):23-33. doi: 10.1111/j.1399-0012.2011.01411.x. Epub 2011 Feb 16. PMID 21323736
- [Background] Bellin MD, Kandaswamy R, Parkey J, Zhang HJ, Liu B, Ihm SH, Ansite JD, Witson J, Bansal-Pakala P, Balamurugan AN, Papas KK, Sutherland DE, Moran A, Hering BJ. Prolonged insulin independence after islet allotransplants in recipients with type 1 diabetes. Am J Transplant. 2008 Nov;8(11):2463-70. doi: 10.1111/j.1600-6143.2008.02404.x. Epub 2008 Sep 19. PMID 18808408
- [Background] Badet L, Benhamou PY, Wojtusciszyn A, Baertschiger R, Milliat-Guittard L, Kessler L, Penfornis A, Thivolet C, Renard E, Bosco D, Morel P, Morelon E, Bayle F, Colin C, Berney T; GRAGIL Group. Expectations and strategies regarding islet transplantation: metabolic data from the GRAGIL 2 trial. Transplantation. 2007 Jul 15;84(1):89-96. doi: 10.1097/01.tp.0000268511.64428.d8. PMID 17627243
- [Derived] Lablanche S, David-Tchouda S, Margier J, Schir E, Wojtusciszyn A, Borot S, Kessler L, Morelon E, Thivolet C, Pattou F, Vantyghem MC, Berney T, Benhamou PY. Randomised, prospective, medico-economic nationwide French study of islet transplantation in patients with severely unstable type 1 diabetes: the STABILOT study protocol. BMJ Open. 2017 Feb 20;7(2):e013434. doi: 10.1136/bmjopen-2016-013434. PMID 28219959